CLINICAL TRIAL: NCT00973830
Title: The Missouri Health Literacy and Diabetes Communication Initiative
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NU0923013
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Diabetes Knowledge
Keywords: Changes in HbA1c

ARMS (3):
- Carve-In (Experimental): Patients in this arm are given the Diabetes Guide and engage in six sessions of brief counseling with a nurse or medical assistant from their clinic. Counseling focuses on behavioral changes patients can make to improve their diabetes.
  Interventions: Other: Diabetes Guide and Brief Counseling
- Carve-Out (Experimental): Patients in this arm are given the Diabetes Guide and engage in six sessions of brief counseling over-the-phone with a diabetes health educator stationed in Chicago, IL. Counseling focuses on behavioral changes patients can make to improve their diabetes.
  Interventions: Other: Diabetes Guide and Brief Counseling
- Control (No Intervention): Patients in this arm receive standard care. They receive no Diabetes Guide or brief counseling sessions

INTERVENTIONS:
Other: Diabetes Guide and Brief Counseling — If in one of the intervention arms, patients will receive a Diabetes Guide (a patient-friendly guide to help patients make healthy changes to improve their diabetes). The Diabetes Guide includes a brief counseling component, to be conducted with clinic staff (Carve-In) or an outside diabetes educator (Carve-Out).
  Arms: Carve-In; Carve-Out

SUMMARY:
Objective: to evaluate the efficacy of the American College of Physicians Foundation (ACPF) Diabetes Guide (Living with Diabetes: An Everyday Guide for You and Your Family) to improve diabetes self-management.

Study Sites: Nine Federally-qualified health centers or safety-net clinics at three sites in Missouri. Sites are urban (St. Louis), midsize (Columbia) and rural (Kirksville). Three FQHCs or safety net clinics are located at each of the sites.

Methods Overview and Design: A randomized controlled trial will be conducted. Patients will be recruited from identified health centers. As the intervention itself is directed to the clinic and not patient, the clinics will be randomly assigned to either 1) usual care (no treatment), 2) "Carve-In" - patients receive the Diabetes Guide and clinic staff follow-up and work with patients to create and complete action plans or 3)"Carve-Out" - patients receive the Diabetes Guide and a diabetes educator in Chicago follows up and works with patients to create and complete action plans. Recruited subjects will be administered a baseline assessment, and 3-month and 1-year follow-up assessments.

Sample: The investigators will recruit a total of 1,080 patients (n=120 per clinic) anticipating 80 percent retention through both follow-up assessments (final estimated number of patients = 720). Eligibility to participate will be defined as patients 1) ages 30 and older (to better represent disease distribution), 2) English or Spanish-speaking, 3) a confirmed (by chart) diagnosis of uncontrolled diabetes (HBA1c 7.0 or more).

ELIGIBILITY:
Inclusion Criteria:

* Uncontrolled diabetes patients (defined as HbA1c 6.0 or greater).
* 25 years or older
* English or Spanish speaking

Exclusion Criteria:

* Uncorrectable hearing or visual impairment
* Moderate to severe cognitive deficits

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 2008-08; Primary Completion 2010-04 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Diabetes knowledge | 3 months, 1 year

SECONDARY OUTCOMES:
Change in HbA1c reading | 3 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michael S. Wolf, PhD, MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States